CLINICAL TRIAL: NCT03394079
Title: A Prospective, Open Label, Multi-center, Dual Arm, Randomized, Pragmatic Trial : Optical Coherence Tomography Versus Intravascular Ultrasound Guided Percutaneous Coronary Intervention
Brief Title: Optical Coherence Tomography Versus Intravascular Ultrasound Guided Percutaneous Coronary Intervention
Acronym: OCTIVUS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, Professor, Division of Cardiology, Division of Cardiology, Asan Medical Center, University of Ulsan, College of Medicine, Seoul, South Korea, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMCCV2017-10
Record Dates: First submitted 2017-12-25; First posted 2018-01-09 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Coronary Vessels
Keywords: OCT; IVUS; PCI

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OCT-guided (Experimental)
  Interventions: Procedure: PCI
- IVUS-guided (Active Comparator)
  Interventions: Procedure: PCI

INTERVENTIONS:
Procedure: PCI — Percutaneous Coronary Intervention

SUMMARY:
The primary aim of this study is to compare the clinical efficacy and safety of OCT-guided(optical coherence tomography (OCT)-guided) and IVUS-guided(Intravascular ultrasound (IVUS)-guided) strategies in patients undergoing Percutaneous coronary intervention (PCI) with contemporary drug-eluting stents (DES) or drug-coated balloons (only for in-stent restenosis) for significant obstructive Coronary artery disease (CAD).

The investigators hypothesize that OCT-guided PCI is non-inferior to IVUS-guided PCI with respect to primary end point of target-vessel failure (cardiac death, target-vessel myocardial infarction [MI], or ischemia-driven target-vessel revascularization [TVR]) at 1 year after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Men or women at least 19 years of age
* Subjects with obstructive CAD undergoing PCI with contemporary DES or drug-coated balloons (only for in-stent restenosis) under intracoronary imaging guidance.
* The patient or guardian agrees to the study protocol and the schedule of clinical follow-up and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site.

Exclusion Criteria:

* ST-elevation myocardial infarction
* Severe renal dysfunction (eGFR <30 ml/min/1.73 m2 or serum creatinine level >1.5 mg/dl), unless patient is on renal replacement therapy.
* Cardiogenic shock or decompensated heart failure with severe LV dysfunction (LVEF) < 30%
* Life expectancy < 1 year for any non-cardiac or cardiac causes
* Any lesion characteristics resulting in the expected inability to deliver the IVUS or OCT catheter to the lesion pre- and post-PCI (eg, moderate or severe vessel calcification or tortuosity)
* Any clinically significant abnormality identified at the screening visit, physical examination, laboratory tests, or electrocardiogram which, in the judgment of the Investigator, would preclude safe completion of the study
* Unwillingness or inability to comply with the procedures described in this protocol

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2008 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Rate of target vessel failure | 1 year
  A composite of cardiac death, target-vessel MI or ischemia-driven TVR) at 1 year after randomization.
  A composite endpoint is an endpoint that is a combination of multiple clinical endpoints. An event is considered to have occurred if any one of several different events is observed.

SECONDARY OUTCOMES:
Rate of cardiac Death | 1, and 5 years
Rate of target vessel myocardial infarction | 1, and 5 years
Rate of ischemia-driven target vessel revascularization | 1, and 5 years
Rate of death | 1, and 5 years
  cardiac, vascular, non-cardiovascular death
Rate of myocardial infarction | 1, and 5 years
  periprocedural or spontaneous, Q-wave or non-Q-wave.
Rate of stent thrombosis | 1, and 5 years
  Stent thrombosis is defined according to according to the definite or probable criteria of the Academic Research Consortium.
Rate of stroke | 1, and 5 years
  Stroke is defined as focal loss of neurologic function caused by an ischemic or hemorrhagic event, with residual symptoms lasting at least 24 hours or leading to death.
Rate of repeat revascularization | 1, and 5 years
  Any, target-lesion or non-target-lesion, target-vessel or non-target-vessel, ischemia-driven or non-ischemia-driven.
Rate of any hospitalization | 1, and 5 years
  Cardiac or non-cardiac causes.
Rate of bleeding events | 1, and 5 years
  Life-threatening or disabling, major bleeding, or minor.
  Bleeding events are assessed according to the Bleeding Academic Research Consortium (BARC) criteria.
Rate of target-lesion failure | 1, and 5 years
  Cardiac death, target-vessel myocardial infarction or ischemia-driven target-lesion revascularization
Rate of contrast-induced acute kidney injury | 3 days
  Contrast-induced nephropathy is defined as either a greater than 25% increase of serum creatinine or an absolute increase in serum creatinine of 0.5 mg/dl within 72 hours after PCI.
Rate of procedural complications requiring active intervention that were related to PCI or intracoronary imaging devices | 1 day
  Procedural complications (e.g., angiographic dissection of at least type B, coronary perforation, vasospasm, thrombus formation, air embolization, slow flow or no reflow, distal embolization, acute closure, ventricular arrhythmia, cardiac tamponade, or cardiogenic shock) requiring active interventions (prolonged balloon inflations, additional stenting required, thrombus aspiration, pericardiocentesis, cardioversion, or use of mechanical circulatory support devices), which are related to PCI procedures or intravascular imaging evaluation.
Rate of angiographic or imaging-based device success | 1 day
  Patient- or lesion-level analysis.
  Angiographic device success is defined as successful PCI at the intended target-lesion with final in-stent residual stenosis of less than 30% by quantitative coronary angiography (QCA). Imaging-based device success is defined as successful PCI at the intended target-lesion, which fulfills the optimal criterial for stent implantation by IVUS or OCT.

CONTACTS AND LOCATIONS:
Overall Officials: Duk-woo Park, MD, Principal Investigator — Professor, Division of Cardiology, Division of Cardiology, Asan Medical Center, University of Ulsan, College of Medicine, Seoul, South Korea
Locations (9):
- South Korea (9):
  - Keimyung University Dongsan Medical Center, Daegu
  - Konyang University Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Pusan National University Hospital, Pusan
  - Asan Medical Hospital, Seoul
  - Chung-Ang university hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Kyung hee university hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim H, Kang DY, Ahn JM, Kim HJ, Hur SH, Cho YK, Lee CH, Hong SJ, Kim SW, Won H, Oh JH, Hong YJ, Yoon YH, Park SJ, Park DW; OCTIVUS Investigators. Proportion and Clinical Impact of Stent Optimization During Imaging-Guided Percutaneous Coronary Intervention: The OCTIVUS Trial. JACC Cardiovasc Interv. 2025 May 12;18(9):1089-1099. doi: 10.1016/j.jcin.2025.01.436. Epub 2025 Apr 23. PMID 40272346
- [Derived] Kang DY, Ahn JM, Yun SC, Hur SH, Cho YK, Lee CH, Hong SJ, Lim S, Kim SW, Won H, Oh JH, Choe JC, Hong YJ, Yoon YH, Kim H, Choi Y, Lee J, Yoon YW, Kim SJ, Bae JH, Park SJ, Park DW; OCTIVUS Investigators. Guiding Intervention for Complex Coronary Lesions by Optical Coherence Tomography or Intravascular Ultrasound. J Am Coll Cardiol. 2024 Jan 23;83(3):401-413. doi: 10.1016/j.jacc.2023.10.017. Epub 2023 Oct 23. PMID 37879490
- [Derived] Kang DY, Ahn JM, Yun SC, Hur SH, Cho YK, Lee CH, Hong SJ, Lim S, Kim SW, Won H, Oh JH, Choe JC, Hong YJ, Yoon YH, Kim H, Choi Y, Lee J, Yoon YW, Kim SJ, Bae JH, Park DW, Park SJ; OCTIVUS Investigators. Optical Coherence Tomography-Guided or Intravascular Ultrasound-Guided Percutaneous Coronary Intervention: The OCTIVUS Randomized Clinical Trial. Circulation. 2023 Oct 17;148(16):1195-1206. doi: 10.1161/CIRCULATIONAHA.123.066429. Epub 2023 Aug 27. PMID 37634092
- [Derived] Kang DY, Ahn JM, Park H, Lee PH, Kang SJ, Lee SW, Kim YH, Park SW, Kim SW, Hur SH, Cho YK, Lee CH, Hong SJ, Hong YJ, Yoon YW, Kim SJ, Bae JH, Oh JH, Park DW, Park SJ. Comparison of optical coherence tomography-guided versus intravascular ultrasound-guided percutaneous coronary intervention: Rationale and design of a randomized, controlled OCTIVUS trial. Am Heart J. 2020 Oct;228:72-80. doi: 10.1016/j.ahj.2020.08.003. Epub 2020 Aug 8. PMID 32871327